CLINICAL TRIAL: NCT06716346
Title: Investigation of Posture, Postural Stability and Core Endurance in Adults with Forward Head Posture: a Controlled Study
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2024/19-15
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Forward Head Posture
Keywords: forward head posture; postural stability; balance; core; endurans

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Forward head posture group: -Craniovertebral angle <50
- control: -Craniovertebral angle >50

SUMMARY:
Forward head posture (FHP) is defined as the position in which the head is in front of the shoulder and is one of the most common musculoskeletal problems caused by increasing computer and smartphone use. The aim of this study is to compare the posture, postural stability and core endurance of participants with normal posture and participants with FHP.

DETAILED DESCRIPTION:
Forward head posture (FHP) is defined as the position in which the head is in front of the shoulder and is one of the most common musculoskeletal problems caused by increasing computer and smartphone use. FHP affects the muscle functions in the neck and thoracic region, reduces the expansion of the rib cage, diaphragm activation and strength with the kyphotic posture it causes, and causes a restrictive pulmonary disorder. In addition, FHP causes various postural alignment disorders in the body, leading to weakening of the core region and affecting postural stability. Posture analysis, postural stability and core endurance tests will be applied to the participants. The aim of this study is to compare the posture, postural stability and core endurance of participants with normal posture and participants with FHP.

ELIGIBILITY:
Inclusion Criteria:

-18-35 years

Exclusion Criteria:

* Diagnosed respiratory, neurological, orthopaedic, psychiatric or cardiac problems
* Pregnancy or breastfeeding
* Having a history of neck trauma
* Having undergone spinal surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with a CVA of 50 degrees and less than 50 degrees will be included in the head forward posture group, and participants with a CVA above 50 degrees will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
postur | Baseline
  A digital camera will be used to assess head and neck posture in the standing position.
Postural stability | Baseline
  Postural stability will be assessed in the bipedal position with eyes open and closed and in the unipedal position with eyes open. All tests will be measured using a force plate platform.

SECONDARY OUTCOMES:
Core endurance | Baseline
  Core endurance is assessed using the trunk flexor test, trunk extensor test and side bridge test. All assessments are carried out during the time the individual is able to remain in bed.

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Demirtaş, Msc., Principal Investigator — Niğde Ömer Halisdemir Üniversitesi
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided